CLINICAL TRIAL: NCT00003681
Title: Phase II Multicenter Study of Amifostine in Patients With Myelodysplastic Syndromes at Relatively Low Risk of Developing Acute Leukemia
Brief Title: Amifostine With or Without Epoetin Alfa in Treating Patients With Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066783; EORTC-06975
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2000-07

CONDITIONS: Anemia; Myelodysplastic Syndromes
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; anemia
MeSH Terms: conditions — Anemia; Myelodysplastic Syndromes; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts | interventions — Epoetin Alfa; Amifostine

INTERVENTIONS:
Biological: epoetin alfa
Drug: amifostine trihydrate

SUMMARY:
RATIONALE: Amifostine may improve blood counts in patients with myelodysplastic syndrome. Epoetin alfa may stimulate red blood cell production and be an effective treatment for anemia in patients with myelodysplastic syndrome.

PURPOSE: Phase II trial to study the effectiveness of amifostine with or without epoetin alfa in treating patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effect of amifostine alone and in combination with epoetin alfa on bone marrow progenitor cells and number of blast cells, blood leukocyte counts, reticulocytes, hemoglobin level, and platelet counts as well as peripheral blood and bone marrow blast cell count in patients with myelodysplastic syndromes at a low risk of developing acute leukemia. II. Determine partial or complete response and duration of response in this patient population. III. Characterize the subjective and objective toxicity of amifostine in these patients.

OUTLINE: This is a multicenter study. Patients receive amifostine IV 3 times per week for 3 weeks followed by 1 week of rest. Response is assessed after 2 courses of therapy. Treatment continues in the absence of disease progression. Patients with complete response receive 1 additional course. Patients with partial response or stable disease are stratified into 2 groups: Group 1: Patients with hemoglobin of at least 10 g/dL without transfusion receive 2 additional courses of amifostine alone. Group 2: Patients with hemoglobin less than 10 g/dL, or who are transfusion dependent, receive 2 additional courses of amifostine in combination with epoetin alfa subcutaneously 3 times per week. Both groups are reevaluated after these 2 additional courses. Treatment may then continue at the discretion of the treating physician. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 27-50 patients will be accrued to this study within 1.3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Confirmed diagnosis of good or intermediate prognosis myelodysplasia of one of the following types: Refractory anemia Refractory anemia with ringed sideroblasts Refractory anemia with excess blasts with no greater than 10% bone marrow blasts No complex abnormalities or involvement of chromosome 7

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: At least 3 months Hematopoietic: Hemoglobin no greater than 10 g/dL OR Transfusion requirement of at least 2 packs RBC per month AND/OR Platelet count no greater than 50,000/mm3 AND/OR Neutrophil count no greater than 1,000/mm3 Hepatic: Bilirubin no greater than 2.5 times upper limit of normal (ULN) SGPT/ALT no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No severe cardiac dysfunction (CTC-NCIC grade III or IV) Pulmonary: No severe pulmonary dysfunction Neurologic: No history of CNS disturbances Other: No current or recent history of allergies No other nonmalignant systemic disease Not pregnant or nursing No active uncontrolled infections Must have cytogenetics done within the past 4 months

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 2 months since prior growth factors or biological response modifiers for myelodysplastic syndrome except for supportive care No other concurrent hematopoietic growth factors Chemotherapy: At least 2 months since other prior chemotherapy for myelodysplastic syndrome Endocrine therapy: No concurrent glucocorticoids No concurrent androgens Radiotherapy: Not specified Surgery: Not specified Other: No concurrent vitamin A or D derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 1998-08

CONTACTS AND LOCATIONS:
Overall Officials: Roel Willemze, MD, PhD, Study Chair — Leiden University Medical Center
Locations (12):
- Universitaetsklinik, Innsbruck, Austria
- Belgium (4):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - A.Z. St. Jan, Bruges
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Universitair Ziekenhuis Antwerpen, Edegem
- Czechia (3):
  - University Hospital - Olomouc, Olomouc
  - Institute of Hematology and Blood Transfusion, Prague
  - Onkologicka Klinka A Onkologicka Lab, Prague (Praha)
- Leiden University Medical Center, Leiden, Netherlands
- Hospital Escolar San Joao, Porto, Portugal
- Institute of Hematology & Transfusiology, University Hospital, Bratislava, Slovakia
- University Hospital, Basel, Switzerland